CLINICAL TRIAL: NCT01340651
Title: An Open-label Assessment of Once-daily Dosing of a Sustained Release (SR) Formulation of INCB018424 in Patients With Primary Myelofibrosis, Post-essential Thrombocythemia Myelofibrosis, and Post-polycythemia Vera Myelofibrosis
Brief Title: Study of Ruxolitinib (INCB018424) Sustained Release Formulation in Myelofibrosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18424-260
Record Dates: First submitted 2011-04-21; First posted 2011-04-22 (Estimated); Results first posted 2013-09-25 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2013-12

CONDITIONS: Myelofibrosis
Keywords: myelofibrosis; myeloproliferative neoplasms; PMF; PET-MF; PPV-MF
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ruxolitinib 25 mg SR/10, 15, or 20 mg IR (Experimental): Participants began administration with 25 mg ruxolitinib sustained release (SR) once daily (QD). After 8 weeks, if there was inadequate efficacy, the dose level could be titrated to 50 mg SR QD or 25 mg SR every other day (QOD) alternating with 50 mg SR QOD. At Week 16, participants transitioned to ruxolitinib 10, 15, or 20 mg immediate release (IR) orally twice daily. Participants who continued to demonstrate benefit in the opinion of the investigator could remain on ruxolitinib IR until the last participant completed Week 36 or the commercial availability of ruxolitinib IR, whichever was earlier; the dose received was based on platelet counts at the time of transition.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib was supplied as SR and IR formulated tablets.
  Other Names: INCB018424

SUMMARY:
The purpose of this study is to determine the safety and tolerability of ruxolitinib (INCB018424) sustained release (SR) formulation in participants with primary myelofibrosis (PMF), post-polycythemia vera MF (PPV-MF), and post-essential thrombocythemia MF (PET-MF).

DETAILED DESCRIPTION:
The study will enroll approximately 40 participants with PMF, PPV-MF or PET-MF. Participants will take ruxolitinib SR once daily for 16 consecutive weeks and then transition to a comparable twice daily dose regimen of ruxolitinib using the immediate release (IR) tablets which have been under investigation in controlled Phase 1, 2, and 3 clinical trials.

Participants receiving benefit from treatment with ruxolitinib may continue further participation with IR tablets up to the time when the last participant completed Week 36 or the commercial availability of ruxolitinib IR, whichever was earlier. Follow-up will occur at least 30 days following the last dose of ruxolitinib.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years of age or older.
* Participants must be diagnosed with primary myelofibrosis (PMF), post-essential thrombocythemia myelofibrosis (PPV-MF), or post-polycythemia vera myelofibrosis (PET-MF).
* Participants with myelofibrosis requiring therapy must be classified as high risk (3 or more prognostic factors), intermediate risk level 2 (2 prognostic factors), or intermediate risk level 1 (1 prognostic factor)defined by International Working Group for Myelofibrosis Research and Treatment (IWG-MRT).
* Participants must have a palpable spleen measuring 5 cm or greater below the costal margin.

Exclusion Criteria:

* Participants with a life expectancy of less than 6 months.
* Participants of childbearing potential who are unwilling to take appropriate precautions to avoid pregnancy or fathering a child.
* Participants with inadequate bone marrow reserve.
* Participants with history of platelet counts < 50,000/μL, platelet transfusion(s), or an absolute neutrophil count < 500/μL in the month prior to Screening.
* Participants with inadequate liver or renal function at Screening and Baseline visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Scottsdale, Arizona
  - Winter Park, Florida
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Ruxolitinib: Participants began administration with 25 mg ruxolitinib sustained release (SR) once daily (QD). After 8 weeks, if there was inadequate efficacy, the dose level could be titrated to 50 mg SR QD or 25 mg SR every other day (QOD) alternating with 50 mg SR QOD. At Week 16, participants transitioned to ruxolitinib 10, 15, or 20 mg immediate release (IR) orally twice daily up to when the last participant completed Week 36 or the commercial availability of ruxolitinib IR, whichever was earlier; the dose received was based on platelet counts at the time of transition.
Period: Overall Study
Arm/Group | Ruxolitinib
Started | 41
Completed | 24
Not Completed | 17
Not completed — Adverse Event | 3
Not completed — Consent Withdrawn | 2
Not completed — Commercial Supply per Sponsor | 12

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All enrolled participants.
Groups:
- Ruxolitinib: Participants began administration with 25 mg ruxolitinib sustained release (SR) once daily (QD). After 8 weeks, if there was inadequate efficacy, the dose level could be titrated to 50 mg SR QD or 25 mg SR every other day (QOD) alternating with 50 mg SR QOD.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (7.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event From Baseline Through Week 16
Time Frame: Baseline to Week 16
Population: Safety population: All enrolled participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 41
Percentage of participants | 78.0

2. Primary Outcome: Overall Response (OR) at Week 16
Description: The investigator graded OR according to the International Working Group for Myelofibrosis Research and Therapy criteria for treatment response. As bone marrow biopsies were not taken after baseline, the best achievable response was clinical improvement which required 1 of the following in the absence of progressive disease (PD): (1) A ≥ 2 g/dL increase in hemoglobin level or (2) either a palpable ≥ 50% reduction of splenomegaly of a spleen ≥ 10 cm at baseline or a spleen palpable at > 5 cm at baseline becoming not palpable. PD required 1 of the following: (1) Progressive splenomegaly defined by the appearance of previously absent splenomegaly that was palpable at > 5 cm below the left costal margin or a ≥ 100% increase in palpable distance for baseline splenomegaly of 5-10 cm or a ≥ 50% increase in palpable distance for baseline splenomegaly of > 10 cm or (2) an increase in peripheral blood blast percentage to ≥ 20% that lasted for ≥ 8 weeks. Stable disease: None of the above.
Time Frame: Baseline to Week 16
Population: Intent-to-treat population: All enrolled participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 41
Percentage of participants
  Clinical improvement | 17.1
  Stable disease | 80.5
  Progressive disease | 2.4

3. Secondary Outcome: Change From Baseline in Spleen Volume at Week 16
Description: Spleen volume was measured by magnetic resonance imaging (or by computed tomography [CT] in applicable participants). Scans were read by a central reader. Spleen volume was obtained by outlining the circumference of the organ and determining the volume using the validated technique of least squares.
Time Frame: Baseline to Week 16
Population: Intent-to-treat population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 40
Percentage change | -22.3 (20.79)

4. Secondary Outcome: Change From Baseline in Spleen Length at Week 16
Description: Spleen length was measured in centimeters by palpation.
Time Frame: Baseline to Week 16
Population: Intent-to-treat population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 38
Percentage change | -29.6 (34.38)

5. Secondary Outcome: Percentage of Participants With ≥ 35% Reduction in Spleen Volume at Week 16 From Baseline
Description: as for outcome 3
Time Frame: Baseline to Week 16
Population: Intent-to-treat population: All enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 41
Percentage of participants | 26.8 [14.2 to 42.9]

6. Secondary Outcome: Change From Baseline in the Total Symptom Score at Week 16
Description: Symptoms of myelofibrosis were assessed using the modified Myelofibrosis Symptom Assessment Form v2.0 diary that was to be completed by participants each night. The 7 symptoms (night sweats, itchiness, abdominal pain, pain under the ribs on left side, feeling of fullness [early satiety], bone/muscle pain, inactivity) were each rated on a scale from 0 (absent) to 10 (worst imaginable). The total symptom score was the sum of 6 of the 7 symptoms (inactivity was not included) and ranged from 0 to 60. A lower score indicated fewer symptoms. A negative change score indicated improvement.
Time Frame: Baseline to Week 16
Population: Intent-to-treat population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 38
Percentage change | -50.4 (31.16)

7. Secondary Outcome: Percentage of Participants With a ≥ 50% Reduction From Baseline in the Total Symptom Score at Week 16
Description: Symptoms of myelofibrosis were assessed using the modified Myelofibrosis Symptom Assessment Form v2.0 diary that was to be completed by participants each night. The 7 symptoms (night sweats, itchiness, abdominal pain, pain under the ribs on left side, feeling of fullness [early satiety], bone/muscle pain, inactivity) were each rated on a scale from 0 (absent) to 10 (worst imaginable). The total symptom score was the sum of 6 of the 7 symptoms (inactivity was not included) and ranged from 0 to 60. A lower score indicated fewer symptoms.
Time Frame: Baseline to Week 16
Population: Intent-to-treat population: All enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 41
Percentage of participants | 43.9 [28.5 to 60.3]

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ruxolitinib 25 mg SR on Day 1
Description: Blood samples were collected prior to and at 0.5, 1, 2, 3, 4, 6, and 9 hours after administration of ruxolitinib 25 mg SR on Day 1 of the study. The concentration of ruxolitinib was determined in plasma samples by a validated LC/MS/MS assay. Standard non-compartmental pharmacokinetic methods were used to analyze the ruxolitinib plasma concentration data using WinNonlin® version 6.0.0 (Pharsight Corporation, Mountain View, CA). Cmax was taken directly from the observed plasma concentration data.
Time Frame: Day 1
Population: Pharmacokinetic evaluable participants: All enrolled participants who received at least 1 dose of study medication and provided at least 1 plasma sample.
Measure: Mean (Standard Deviation); unit: nM
Groups:
- Ruxolitinib: Participants began administration with 25 mg ruxolitinib sustained release (SR) once daily (QD).
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 41
nM | 319 (119)

9. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Ruxolitinib 25 mg SR on Day 1
Description: Blood samples were collected prior to and at 0.5, 1, 2, 3, 4, 6, and 9 hours after administration of ruxolitinib 25 mg SR on Day 1 of the study. The concentration of ruxolitinib was determined in plasma samples by a validated LC/MS/MS assay. Standard noncompartmental pharmacokinetic methods were used to analyze the ruxolitinib plasma concentration data using WinNonlin® version 6.0.0 (Pharsight Corporation, Mountain View, CA). Tmax was taken directly from the observed plasma concentration data.
Time Frame: Day 1
Population: as for outcome 8
Measure: Median (Full Range); unit: h
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 41
h | 2.0 [0.5 to 8.8]

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) of Ruxolitinib 25 mg SR on Day 1
Description: Blood samples were collected prior to and at 0.5, 1, 2, 3, 4, 6, and 9 hours after administration of ruxolitinib 25 mg SR on Day 1 of the study. The concentration of ruxolitinib was determined in plasma samples by a validated LC/MS/MS assay. The area under the plasma concentration-time curve (AUC) was derived from the plasma concentrations using a non-compartmental method and computed using the linear trapezoidal rule for increasing concentrations and the log-trapezoidal rule for decreasing concentrations with the software WinNonlin® version 6.0.0 (Pharsight Corporation, Mountain View, CA).
Time Frame: Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nM*h
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 41
nM*h | 1550 (647)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline through the end of the study
Description: Safety population: All enrolled participants who took at least 1 dose of study drug.
Groups:
- Ruxolitinib - Weeks 1-16: Participants began administration with 25 mg ruxolitinib sustained release (SR) once daily (QD). After 8 weeks, if there was inadequate efficacy, the dose level could be titrated to 50 mg SR QD or 25 mg SR every other day (QOD) alternating with 50 mg SR QOD.
- Ruxolitinib - After Week 16: At Week 16, participants transitioned to ruxolitinib 10, 15, or 20 mg immediate release (IR) orally twice daily up to when the last participant completed Week 36 or the commercial availability of ruxolitinib IR, whichever was earlier; the dose received was based on platelet counts at the time of transition.
Arm/Group | Ruxolitinib - Weeks 1-16 | Ruxolitinib - After Week 16
Serious Adverse Events (participants affected / at risk) | 6/41 | 9/41
Other Adverse Events (participants affected / at risk) | 27/41 | 9/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib - Weeks 1-16 (N=41) | Ruxolitinib - After Week 16 (N=41)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Generalized edema (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Prostate infection (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib - Weeks 1-16 (N=41) | Ruxolitinib - After Week 16 (N=41)
Diarrhoea (Gastrointestinal disorders) | 8 | 4
Nausea (Gastrointestinal disorders) | 3 | 0
Oedema peripheral (General disorders) | 7 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Asthenia (General disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Sinusitis (Infections and infestations) | 3 | 0
Platelet count decreased (Investigations) | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least thirty (30) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.